CLINICAL TRIAL: NCT00317577
Title: A Multicenter, Double-Masked, 2-Arm Parallel Group Study Comparing the Effect of Brimonidine 0.2% Versus Timolol 0.5% on Visual Field Stability in Patients With Low-Pressure Glaucoma
Brief Title: Study of Medical Treatment of Low-Pressure (Normal Tension) Glaucoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chicago Center for Vision Research (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCVR-0020
Record Dates: First submitted 2006-04-23; First posted 2006-04-25 (Estimated); Last update posted 2006-04-25 (Estimated); Status verified 2006-04

CONDITIONS: Glaucoma, Open Angle
Keywords: Low-pressure glaucoma; Normal tension glaucoma; Neuroprotection; Brimonidine; Visual field progression
MeSH Terms: conditions — Glaucoma, Open-Angle; Low Tension Glaucoma | interventions — Brimonidine Tartrate, Timolol Maleate Drug Combination

INTERVENTIONS:
Drug: brimonidine, timolol

SUMMARY:
Low-pressure (normal tension) glaucoma is a type of open-angle glaucoma resulting in damage to the optic nerve and abnormalities of the visual field. Eye (intraocular) pressure in this type of glaucoma is not higher than that usually considered to be normal (less than 21 mmHg) for the eye. The present treatment of low-pressure glaucoma is also directed to lowering the "normal" eye pressure. Both medications in this study, brimonidine and timolol, lower eye pressure.

Laboratory research over the past decade indicates the potential to treat glaucoma not only by lowering eye pressure, but with treatments aimed at the damage occurring at the optic nerve. One group of drugs, selective alpha2-adrenergic agonists, have been shown in laboratory animals to protect against the effects of nerve damage following local stroke. Brimonidine, one of the medications in the current study, is a selective alpha2-adrenergic agonist which protects against damage to optic nerve in animal models of glaucoma..

The hypothesis of the present study is that brimonidine eye drops provide protection to the damaged optic nerve independent of lowering eye pressure in patients with low-pressure glaucoma. This will be determined by (1) measuring eye pressure, (2) performing visual field examinations, and (3) examination of the optic nerve.

DETAILED DESCRIPTION:
The term glaucoma describes a specific pattern of optic nerve head and visual field damage caused by a number of different diseases of the eye, most (but not all) of which are associated with an elevated eye pressure. Glaucoma is currently considered to be a progressive neurodegenerative disorder. Low-pressure glaucoma (LPG) is a type of open-angle glaucoma (OAG) with progressive visual field and optic nerve damage despite an untreated eye pressure in the statistically normal (mean 15.9, SD 2.9 mmHg) range, usually less than 21 mmHg. Therefore, in this condition, pressure-independent mechanisms (e.g., vascular or structural defects of the optic nerve) may be the main, if not the sole, cause of the optic neuropathy. LPG represents 6.7% to 68.3% of all OAGs.

Current glaucoma treatment is directed to lowering eye pressure using medical therapy (eye drops), laser treatment, and/or surgery, to a level that stops progressive optic nerve damage. The efficacy of lowering eye pressure in LPG has been reported. Both protocol medical treatments, brimonidine and timolol, show similar efficacy to lower eye pressure.

Laboratory research over the past decade indicates the potential to manage glaucoma not only by lowering eye pressure, but with treatment modalities aimed at the damage occurring at the optic nerve. Possible therapies may include agents effective as neuronal protectants to increase or prolong the survival rate of injured retinal ganglion cells. Treatments could also be directed to the rescue of nerve fibers from secondary degeneration, as stimulants to expand dendritic fields, and to promote nerve regeneration or neural transplantation.

Selective α2-adrenergic agonists have been shown to have a neuroprotective effect in animal models of focal cerebral ischemia. Brimonidine is reported to protect the optic nerve and retinal ganglion cells from secondary degeneration following a partial crush lesion to the adult rat optic nerve. One molecular mechanism for this neuroprotection may relate to up-regulation of neuronal survival factors. In rats, systemic α2-adrenergic agonists induce basic fibroblast growth factor mRNA in the retina. Treatment with α2-agonists before and during constant light exposure reduces retinal photoreceptor degeneration in albino rats. Animal studies demonstrate that topical administration of brimonidine results in pharmacologic concentrations of drug in the vitreous (100-170 nM). Therefore, ocular dosing with brimonidine provides a route for drug delivery to the retina in amounts sufficient to bind and activate the α2-adrenoceptor and provide a neuroprotective effect.

The study hypothesis is to evaluate the ability of topical treatment with 0.2% brimonidine, a highly selective α2-adrenergic agonist, to impart neuroprotection to the damaged optic nerve in patients with LPG. Comparison is made to 0.5% timolol, a nonselective β-adrenergic antagonist, without reported neuroprotective properties. Patients will be randomly assigned to twice daily double-masked treatment with one of these drugs. Neuroprotection will be assessed by evaluation of automated static visual fields performed at 4 month intervals for 4 years of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age: 30 years or older.
* Low-pressure glaucoma in at least one eye: untreated IOP < 21 mmHg, glaucomatous field loss on Humphrey 24-2 perimetry, and optic disc cupping.
* Best corrected visual acuity at least 20/40 in at least one eye.
* At least two visual fields within the 6 months prior to enrollment.
* Phakic or pseudophakic (cataract surgery > one year to enrollment) eye.

Exclusion Criteria:

Either eye patient exclusion:

* Past history of confirmed treated or untreated applanation IOP > 21 mmHg.
* Untreated IOP of > 21 mmHg on diurnal curve on Study Day 0.
* Untreated IOP > 4 mmHg difference between the two eyes.
* Extensive field damage: MD > 15 dB or threat fixation in both hemi fields.
* Evidence of exfoliation or pigment dispersion.
* History of angle-closure or occludable gonioscopic anterior chamber angle.
* Prior filtration surgery.
* Prior laser iridotomy.
* Laser trabeculoplasty < 6 months prior enrollment or for an IOP > 21 mmHg.
* History of chronic inflammatory eye diseases (e.g., scleritis, uveitis).
* History or signs of intraocular trauma.
* Severe or potentially progressive retinal disease.
* Any abnormality preventing reliable applanation tonometry.
* History of hypersensitivity to study medications or their components.
* Current use of any ophthalmic, dermatologic or systemic steroid preparation.
* Therapy with another investigational agent within the past 30 days.

Single eye exclusion:

* Cataract surgery within the past year.
* Aphakia.
* Only sighted eye.

Concomitant conditions:

* Resting pulse < 50 beats per minute.
* Unstable or uncontrolled cardiovascular, renal, or pulmonary disease.
* Recent heart attack or stroke.
* Women contemplating pregnancy, who are pregnant or are a nursing mother.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 1998-12; Study Completion 2004-05

PRIMARY OUTCOMES:
To compare changes in automated static visual field decibel values at 4 month intervals over 4 years of monotherapy with either brimonidine or timolol eye drops.

SECONDARY OUTCOMES:
To characterize the intraocular pressure throughout the study period.
To characterize optic disc changes (e.g., cupping and disc hemorrhages) over the 4 years of treatment with brimonidine or timolol.
To follow the safety parameters throughout the study period.
To determine risk factors for visual field progression in low-pressure glaucoma

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Krupin, M.D., Study Chair — Northwestern University Feinberg School of Medicine
Locations (12):
- United States (12):
  - Little Rock Eye Clinic, Little Rock, Arkansas
  - University of Florida, Gainesville, Florida
  - Bascom Palmer Eye Institute, Palm Beach Gardens, Florida
  - University Eye Specialists, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Wheaton Eye Clinic, Wheaton, Illinois
  - Indiana University, Indianapolis, Indiana
  - New York Eye & Ear Infirmary, New York, New York
  - Scheie Eye Institute University of Pennsylvania, Philadelphia, Pennsylvania
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Cullen Eye Institute Baylor University, Houston, Texas

REFERENCES:
- [Background] Krupin T, Liebmann JM, Greenfield DS, Rosenberg LF, Ritch R, Yang JW; Low-Pressure Glaucoma Study Group. The Low-pressure Glaucoma Treatment Study (LoGTS) study design and baseline characteristics of enrolled patients. Ophthalmology. 2005 Mar;112(3):376-85. doi: 10.1016/j.ophtha.2004.10.034. PMID 15745762
- [Derived] Furlanetto RL, De Moraes CG, Teng CC, Liebmann JM, Greenfield DS, Gardiner SK, Ritch R, Krupin T; Low-Pressure Glaucoma Treatment Study Group. Risk factors for optic disc hemorrhage in the low-pressure glaucoma treatment study. Am J Ophthalmol. 2014 May;157(5):945-52. doi: 10.1016/j.ajo.2014.02.009. Epub 2014 Feb 7. PMID 24513094
- [Derived] De Moraes CG, Liebmann JM, Greenfield DS, Gardiner SK, Ritch R, Krupin T; Low-pressure Glaucoma Treatment Study Group. Risk factors for visual field progression in the low-pressure glaucoma treatment study. Am J Ophthalmol. 2012 Oct;154(4):702-11. doi: 10.1016/j.ajo.2012.04.015. Epub 2012 Jul 25. PMID 22835512
- [Derived] Krupin T, Liebmann JM, Greenfield DS, Ritch R, Gardiner S; Low-Pressure Glaucoma Study Group. A randomized trial of brimonidine versus timolol in preserving visual function: results from the Low-Pressure Glaucoma Treatment Study. Am J Ophthalmol. 2011 Apr;151(4):671-81. doi: 10.1016/j.ajo.2010.09.026. Epub 2011 Jan 22. PMID 21257146